CLINICAL TRIAL: NCT07382843
Title: The Study of the Relationship Between Sleep Pattern, Attention Performance, and Heart Rate Variability Among Night Workers.
Brief Title: Melatonin Agonist for Shift-time Workers.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chin-Bin Yeh, MD, PhD, Principal Investigator, Professor, Tri-Service General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C202205038
Record Dates: First submitted 2025-09-03; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Circadian Rhythm Disorders
Keywords: melatonin; chronotype
MeSH Terms: conditions — Chronobiology Disorders | interventions — ramelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ramelteon (Other): comparison of anxiety/depression, insomnia symptoms severity between before and after treatment with 8mg Ramelteon per day for two weeks among shift time workers.
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: Ramelteon — comparison of anxiety/depression, insomnia symptoms severity between before and after treatment with 8mg Ramelteon per day for two weeks among shift time workers.
  Other Names: Rozerem

SUMMARY:
The study of the relationship between sleep pattern, attention performance, and heart rate variability among night workers.

DETAILED DESCRIPTION:
Background: Previous study found that sleeping in the morning or evening pattern might be associated with performance among night workers. Both their sleep quality and circadian rhythm are critical for the performance at night. The study aims to identify the association between sleep pattern and performance among night workers. The effectiveness of interventions either supplement with melatonin for those who not meeting the DSM-5 criteria of Circadian Rhythm Sleep-Wake Disorders, CRSWD and prescription of melatonin agonist ramelteon for those who meet the DSM-5 criteria of CRSWD will be evaluated.

Methods:

The investigators will prescribe melatonin agonist ramelteon for 80 subjects those who agree to participate and meet the DSM-5 diagnostic criteria of this Circadian Rhythm Sleep Wake Disorders. They will receive the assessments including questionnaires and performance measurements before and after prescription with melatonin agonist 8 mg for 2 weeks to investigate the effectiveness of melatonin agonist.

Anticipated outcome: The study will help the understanding the association of sleep pattern and performance among night workers. The effectiveness of either supplement with melatonin and prescription of melatonin agonist will be evaluated. The findings of our study might be implicated in the plans of intervention for better performance for night warriors.

ELIGIBILITY:
Inclusion Criteria:

* The individuals aged 20-55 who are night workers whose working hours more than 4 hours duration between 22:00 to 06:00.
* Meet the DSM-5 diagnostic criteria of this Circadian Rhythm Sleep Wake Disorders.

Exclusion Criteria:

* The individuals could not understand the online questionnaires and is not willing to fill out questionnaires.
* The individual is not willing to have supplement with melatonin.
* Not willing to have prescription with melatonin agonist ramelteon.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index (PSQI） | 2 weeks
  The investigators will measure if the severity improve after using Somn Well XR and Rozerem by the PSQI scale.
  The cutoff score for the cutoff score for the Pittsburgh Sleep Quality Index (PSQI) questionnaire is 5. Higher scores on both questionnaires indicate a greater severity of sleep issues.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | 2 weeks
  The investigators will measure if the severity improve after using Somn Well XR and Rozerem by the BDI scale.
  The cutoff score for the Beck Depression Inventory (BDI) questionnaire is 13. Higher scores on both questionnaires indicate greater severity of depressive and anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Bin Yeh, M.D., Ph.D., Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

DOCUMENTS (1):
  • Study Protocol: Study Protocol_20260126 (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT07382843/Prot_000.pdf